CLINICAL TRIAL: NCT03908164
Title: Optimising the Timing of Whooping Cough Immunisation in MUMs
Acronym: OpTIMUM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Thrasher Research Fund (Other); Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018.0297
Record Dates: First submitted 2019-01-29; First posted 2019-04-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Related; Immunization; Infection; Pertussis
Keywords: Pregnancy; Immunisation; Pertussis
MeSH Terms: conditions — Infections; Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccination at <23+6 gestational weeks (Experimental): Participants will receive a pertussis containing vaccine licensed for use in pregnancy before 23+6 gestational weeks (GW). Although the time period for study group 1 is ≤23+6 no pertussis vaccine will be given in this study at less than 16 GW.
  Interventions: Biological: Pertussis containing vaccine
- Vaccination at 24-27+6 gestational weeks (Experimental): Participants will receive a pertussis containing vaccine licensed for use in pregnancy between 24 and 27+6 gestational weeks.
  Interventions: Biological: Pertussis containing vaccine
- Vaccination at 28-31+6 gestational weeks (Experimental): Participants will receive a pertussis containing vaccine licensed for use in pregnancy between 28 and 31+6 gestational weeks.
  Interventions: Biological: Pertussis containing vaccine

INTERVENTIONS:
Biological: Pertussis containing vaccine — Participants will receive a pertussis containing vaccine licensed for use in pregnancy at one of three time periods.

SUMMARY:
A multicentre study to evaluate the impact of timing of whooping cough (pertussis) vaccination in pregnancy, with participants randomised to receive whooping cough vaccination at one of three time points in pregnancy.

DETAILED DESCRIPTION:
Pertussis is a highly infectious respiratory illness caused by Bordetella pertussis, which characteristically causes paroxysms of coughing with an associated inspiratory 'whoop'. In young infants the clinical presentation can be atypical, is frequently associated with apnoeic episodes and can cause significant morbidity and mortality. Following the introduction of pertussis vaccination into routine infant schedules worldwide there was a significant reduction in the incidence of pertussis. However, recently in a number of countries, despite high vaccine coverage, there has been a resurgence of pertussis disease associated with an increase in infant deaths. Various strategies to control the increasing burden of infant pertussis disease have been considered including cocooning, a strategy in which close contacts of an infant are vaccinated, a neonatal dose of a pertussis containing vaccine, the addition of an adolescent dose to the schedule and vaccination in pregnancy. Of these, the latter has gained most support.

Vaccination in pregnancy is a strategy which relies on effective transport of antibody across the placenta, a process which depends on the antibody available, the gestation of the pregnancy and the health of the placenta. In the case of pertussis, the main aim is to prevent disease in babies (prior to the age of routine vaccination) as they have a higher mortality than any other age group from pertussis disease.

It is now clear that pertussis vaccination in pregnancy can reduce the burden of disease in young infants in the period prior to them being fully immunised, and can do so safely. However, it is not established whether there is an optimal time to vaccinate in pregnancy to ensure maximal protection of the infant. This is reflected in the different guidelines currently in place in different countries: in the UK vaccination is advised from 16 weeks gestation, in Canada from 26 weeks, in the USA from 27 weeks and in Australia from 28 weeks.

While some studies have suggested that vaccination later in pregnancy can achieve higher antibody concentrations in the newborn, others have found earlier vaccination provides improved immunity compared to later vaccination. The significance of this is that if earlier vaccination is shown to be equivalent, there are clear logistical benefits in allowing the widest possible time window in order to maximise the opportunities for pregnant women to be vaccinated and thereby improve vaccine coverage.

When the pertussis vaccination in pregnancy programmes were first implemented, vaccination was recommended in the third trimester (USA 27-36 weeks, UK 28-32 weeks). This decision was based on the hypothesis that vaccination would be most effective if it was timed to allow the peak in maternal antibody levels after vaccination to coincide with the time of most efficient placental transport.

There is a significant lack of agreement on optimal timing of pertussis vaccination in pregnancy due to conflicting data. This is the rationale for this randomised controlled trial.

In this study all participants will receive a pertussis containing vaccine licensed for use in pregnancy. In the UK currently the vaccine used is Boostrix-IPV® manufactured by GlaxoSmithKline. This vaccine contains pertussis toxin (PT) (8 micrograms), filamentous haemagglutinin (FHA) (8 micrograms) and pertactin (PRN) (2.5 micrograms) as well as diphtheria toxoid (not less than 2 international units), tetanus toxoids (not less than 20 international units) and inactivated polio virus types 1-3 (type 1 40 D-antigen unit, type 2 8 D-antigen unit, type 3 32 D-antigen unit). This vaccine will be given at the time period assigned by randomisation. All possible time periods included in the study are within that recommended in the UK as part of routine practice.

Participants will have blood sampling prior to vaccination, 14 days following vaccination and at the time of delivery. At delivery a cord blood sample will also be obtained and an infant sample taken from the infants of participating women at 28-42 days after completion of their primary immunisations.

There is a paucity of information about functional immunity of anti-PT antibody in serum and colostrum/breastmilk following vaccination in pregnancy. We will be investigating this in two exploratory sub-studies. The first of these (investigation of functional immunity of anti-PT antibody in serum) will be performed on samples being performed as part of the main study. For investigation of functional immunity of anti-PT antibody in colostrum and breastmilk we will ask participants at two participating institutions if they are willing to participate in a breastfeeding sub-study if they decide to breastfeed. For participants who take part in this sub-study a sample of colostrum will be obtained within 48 hours of delivery and a further breast milk sample at 14 days and 5 months following delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and not yet having received pertussis vaccination
* Willing and able to comply with study procedures and provide informed consent
* Documentation of a 20-week anomaly scan with no life limiting congenital anomalies identified

Exclusion Criteria:

* Age less than 16 years
* Confirmed or suspected pertussis in previous five years
* Known diagnosis of immune deficiency
* Receiving immunosuppressive medication within six months of enrolment in the study (this does not include inhaled or topical steroids)
* In the opinion of the investigator is unlikely to complete follow up

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Pertussis specific antibody concentration in cord blood of term infants | Delivery of infant
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) from cord blood of term infants. This will be measured using ELISA.

SECONDARY OUTCOMES:
Pertussis specific antibody concentration in cord blood of preterm infants | Delivery of infant
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) from cord blood of preterm infants. This will be measured using ELISA.
Kinetics of antibody response to pertussis vaccination during pregnancy | Prior to vaccination, 14 days following vaccination, delivery
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) in maternal blood prior to vaccination, 14 days following vaccination and at delivery. This will be measured using ELISA.
Placental transfer of antibody | Time of delivery
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) in maternal and cord blood at time of delivery. This will be measured using ELISA.
Impact of repeated vaccination on antibody response in women who have received a pertussis vaccination in a previous pregnancy | Prior to vaccination, 14 days following vaccination and at delivery
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) in maternal blood prior to vaccination, 14 days following vaccination and at delivery. This will be measured using ELISA.
Antibody concentration in infants following primary immunisation schedule | 28-42 days following completion of primary immunisations
  Antibody concentrations against Pertussis Toxin (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) from the infant following primary immunisations. This will be measured using ELISA.

OTHER OUTCOMES:
Functional assays on serum | Samples collected following vaccination, from the cord blood at delivery and in the infants following primary vaccination.
  Serum bactericidal assays will be performed. The bactericidal titre is the last serum dilution where ≥50% killing is observed compared to complement only control. Serum bactericidal assays will be performed and the bactericidal titre will be compared according to the time of vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Heath, Study Chair — St George's, University of London
Locations (1):
- St Georges University Hospital NHS Foundation Trust, Tooting, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvert A, Amirthalingam G, Andrews N, Basude S, Coleman M, Cuthbertson H, England A, Greening V, Hallis B, Johnstone E, Jones CE, Karampatsas K, Khalil A, Le Doare K, Matheson M, Peregrine E, Snape MD, Vatish M, Heath PT; OpTIMUM Study Group. Optimising the timing of whooping cough immunisation in mums (OpTIMUM) through investigating pertussis vaccination in pregnancy: an open-label, equivalence, randomised controlled trial. Lancet Microbe. 2023 May;4(5):e300-e308. doi: 10.1016/S2666-5247(22)00332-9. Epub 2023 Apr 17. PMID 37080224